CLINICAL TRIAL: NCT02726698
Title: Reappraisal of Atrial Fibrillation: Interaction Between HyperCoagulability, Electrical Remodeling, and Vascular Destabilisation in the Progression of Atrial Fibrillation - An Observational Exploratory Study on Pathophysiological Mechanisms of AF Progression and on the Role of LinQ/CareLink Guided Patient Tailored Therapy in Patients With Atrial Fibrillation
Brief Title: Reappraisal of Atrial Fibrillation: Interaction Between HyperCoagulability, Electrical Remodeling, and Vascular Destabilisation in the Progression of Atrial Fibrillation
Acronym: RACE V
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, I.C. Van Gelder, Prof.dr., University Medical Center Groningen
Other Study IDs: NL53561.042.16
Record Dates: First submitted 2016-03-17; First posted 2016-04-04 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to study clinical factors and (blood) biomarkers related to progression of Atrial Fibrillation (AF) in patients diagnosed with self-terminating AF with special reference to hypercoagulability. All patients will be continuously monitored for their atrial rhythm to assess AF progression, either through an implantable loop recorder (Reveal LinQ) or via the atrial lead of a cardiac implantable electronic device (CIED), both in combination with the CareLink home monitoring system. Remote monitoring and interrogation will be installed and used on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* New onset or history of paroxysmal, self-terminating AF documented as:

  * AF on ECG or Holter-recording or loop recorder
  * Subclinical AF detected in implantable cardiac devices (atrial read > 190 beats per minute, lasting > 6 minutes).
* Prior history of self-terminating AF is allowed;
* Able and willing to sign informed consent for the registry;
* Able and willing to undergo implantation of an implantable loop recorder (in patients without a CIED);
* In patients already on oral anticoagulation drugs, the following inclusion criteria need to be met (to allow for safe temporary interruption of anti-thrombotic treatment for coagulation phenotyping):

  * CHA2DS2-VASc score ≤5 (history of Congestive heart failure, Hypertension, Age ≥ 75 years (doubled), Diabetes mellitus,Stroke/transient ischemic attack (doubled), Vascular disease, Age 65-75 years, female Sex);
  * No other indication for oral anticoagulation (e.g. mechanical valve prosthesis);
  * Patient is willing to temporarily stop oral anticoagulation drugs (OAC).

Exclusion Criteria:

* Non-self-terminating, persistent AF;
* Deemed unsuitable or not willing to undergo implantation of loop recorder (in patients without a CIED);
* Refusing to temporarily stop OAC for coagulation phenotyping (in patients already on OAC before inclusion in this study);
* On waiting list for pulmonary vein isolation or expected to be placed on waiting list within one year;
* Expected to start with amiodarone;
* Pregnancy;
* Life expectancy of less than 2.5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal (self-terminating) AF in the cardiology outpatient department, first (heart) aid and pacemaker clinic.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2024-10 (Actual); Study Completion 2024-10 (Actual)

PRIMARY OUTCOMES:
Progression of AF burden | 2.5 years

SECONDARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events | 2.5 years
Change in therapy due to continuous rhythm monitoring with the LinQ/Carelink system | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Harry JGM Crijns, MD, PhD, Principal Investigator — Maastricht University Medical Center; Isabelle C van Gelder, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (9):
- Netherlands (9):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - Amsterdam University Medical Center - AMC, Amsterdam
  - Amsterdam University Medical Center - VU, Amsterdam
  - University Medical Center Groningen, Groningen
  - Martini Hospital, Groningen
  - Ommelander Ziekenhuis, Groningen
  - Laurentius Hospital, Roermond
  - Isala, Zwolle

REFERENCES:
- [Derived] Frausing MHJP, Rienstra M, Kronborg MB, De Melis M, Schotten U, Nielsen JC, Tieleman R, Crijns HJ, Van Gelder IC, Samuel M. Association between circulating biomarkers and atrial fibrillation burden in patients with paroxysmal atrial fibrillation: a subanalysis of the RACE V study. Open Heart. 2025 Sep 30;12(2):e003433. doi: 10.1136/openhrt-2025-003433. PMID 41033708
- [Derived] van Deutekom C, van de Lande ME, Rama R, Nguyen BO, Tieleman RG, Weberndorfer V, Hemels MEW, de Melis M, Schotten U, Linz D, Crijns HJGM, van Gelder IC, Rienstra M; RACE V Investigators. Multimorbidity Is Associated With Symptom Severity and Disease Progression in Patients with Paroxysmal Atrial Fibrillation-Data From the RACE V Study. J Am Heart Assoc. 2025 Mar 4;14(5):e034514. doi: 10.1161/JAHA.123.034514. Epub 2025 Feb 26. PMID 40008502
- [Derived] Koldenhof T, Van Gelder IC, van de Lande ME, Al-Jazairi MIH, Tieleman RG, Rienstra M. High heart rates during paroxysmal atrial fibrillation: continuous rhythm monitoring data of the RACE V study. Heart. 2024 Oct 10;110(21):1250-1253. doi: 10.1136/heartjnl-2024-324376. PMID 39168591
- [Derived] Frausing MHJP, Van De Lande M, Linz D, Crijns HJGM, Tieleman RG, Hemels MEW, De Melis M, Schotten U, Kronborg MB, Nielsen JC, Van Gelder I, Rienstra M. Healthcare utilisation and quality of life according to atrial fibrillation burden, episode frequency and duration. Heart. 2024 Jul 25;110(16):1030-1039. doi: 10.1136/heartjnl-2024-324016. PMID 38944418
- [Derived] van de Lande ME, Rama RS, Koldenhof T, Arita VA, Nguyen BO, van Deutekom C, Weberndorfer V, Crijns HJGM, Hemels MEW, Tieleman RG, de Melis M, Schotten U, Linz D, Van Gelder IC, Rienstra M; RACE V Investigators. Time of onset of atrial fibrillation and atrial fibrillation progression data from the RACE V study. Europace. 2023 May 19;25(5):euad058. doi: 10.1093/europace/euad058. PMID 36967470
- [Derived] Frausing MHJP, Van De Lande ME, Maass AH, Nguyen BO, Hemels MEW, Tieleman RG, Koldenhof T, De Melis M, Linz D, Schotten U, Weberndorfer V, Crijns HJGM, Van Gelder IC, Nielsen JC, Rienstra M. Brady- and tachyarrhythmias detected by continuous rhythm monitoring in paroxysmal atrial fibrillation. Heart. 2023 Aug 11;109(17):1286-1293. doi: 10.1136/heartjnl-2022-322253. PMID 36948572
- [Derived] Artola Arita V, Van De Lande ME, Khalilian Ekrami N, Nguyen BO, Van Melle JM, Geelhoed B, De With RR, Weberndorfer V, Erkuner O, Hillege H, Linz D, Ten Cate H, Spronk HMH, Koldenhof T, Tieleman RG, Schotten U, Crijns HJGM, Van Gelder IC, Rienstra M. Clinical utility of the 4S-AF scheme in predicting progression of atrial fibrillation: data from the RACE V study. Europace. 2023 Apr 15;25(4):1323-1331. doi: 10.1093/europace/euac268. PMID 36857318
- [Derived] Nguyen BO, Weberndorfer V, Crijns HJ, Geelhoed B, Ten Cate H, Spronk H, Kroon A, De With R, Al-Jazairi M, Maass AH, Blaauw Y, Tieleman RG, Hemels MEW, Luermans J, de Groot J, Allaart CP, Elvan A, De Melis M, Scheerder C, van Zonneveld AJ, Schotten U, Linz D, Van Gelder I, Rienstra M. Prevalence and determinants of atrial fibrillation progression in paroxysmal atrial fibrillation. Heart. 2022 Jul 20;109(3):186-94. doi: 10.1136/heartjnl-2022-321027. Online ahead of print. PMID 35858774
- [Derived] De With RR, Artola Arita V, Nguyen BO, Linz D, Ten Cate H, Spronk H, Schotten U, Jan van Zonneveld A, Erkuner O, Bayon MA, Schmidt AS, Luermans JGLM, Crijns HJGM, Van Gelder IC, Rienstra M. Different circulating biomarkers in women and men with paroxysmal atrial fibrillation: results from the AF-RISK and RACE V studies. Europace. 2022 Feb 2;24(2):193-201. doi: 10.1093/europace/euab179. PMID 34329401
- [Derived] De With RR, Erkuner O, Rienstra M, Nguyen BO, Korver FWJ, Linz D, Cate Ten H, Spronk H, Kroon AA, Maass AH, Blaauw Y, Tieleman RG, Hemels MEW, de Groot JR, Elvan A, de Melis M, Scheerder COS, Al-Jazairi MIH, Schotten U, Luermans JGLM, Crijns HJGM, Van Gelder IC; RACE V Investigators. Temporal patterns and short-term progression of paroxysmal atrial fibrillation: data from RACE V. Europace. 2020 Aug 1;22(8):1162-1172. doi: 10.1093/europace/euaa123. PMID 32642768